CLINICAL TRIAL: NCT06923748
Title: Comparison of Two Different Interproximal Cleaning Devices Around Dental Implants: A Randomized Clinical Trial
Brief Title: Comparison of Two Interdental Devices for Peri-Implant Plaque Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Associate Professor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INT001
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis
Keywords: Peri-implant mucositis; Peri-implantitis; Interproximal devices; Prevention
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superfloss (Experimental): Participants in this group will receive an electronic toothbrush combined with Superfloss as the interproximal cleaning aid. Personalized oral hygiene instructions and professional maintenance will be provided throughout the study.
  Interventions: Device: Superfloss
- Interdental Brush (Experimental): Participants in this group will receive an electronic toothbrush combined with interdental brushes for interproximal cleaning. Tailored oral hygiene guidance and professional care will be offered during the follow-up visits.
  Interventions: Device: Interdental brush

INTERVENTIONS:
Device: Superfloss — Use of Superfloss daily as the interproximal cleaning device, combined with an electronic toothbrush, as part of a tailored oral hygiene protocol in patients with peri-implant disease.
  Arms: Superfloss
Device: Interdental brush — Use of interdental brush once daily as the interproximal cleaning device, combined with an electronic toothbrush, within a professional oral hygiene maintenance program for peri-implant disease
  Arms: Interdental Brush

SUMMARY:
This randomized clinical trial aims to compare the efficacy of two interproximal cleaning devices-superfloss and interdental brushes- in patients diagnosed with peri-implant diseases. The study evaluates plaque control and bleeding scores. Patients will be randomly assigned to one of two oral hygiene protocols and will be monitored through clinical examinations and validated questionnaires assessing both clinical and radiographic parameters and patient-reported outcomes.

DETAILED DESCRIPTION:
This single-center, randomized, parallel-arm clinical trial aims to compare the efficacy of superfloss and interdental brushes, used in combination with an electronic toothbrush, in patients with peri-implant diseases. Participants will be randomly assigned to one of two oral hygiene protocols. Clinical assessments will be performed at baseline, 6 weeks, and 3 months, including plaque index, bleeding scores, and probing depth. Radiographic measurements and standardized patient-reported questionnaires (food impaction and oral hygiene self-efficacy) will also be used. The primary outcome is the reduction of plaque and gingival inflammatory scores at implant sites.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Presence of at least one implant loaded for ≥1 year
* Presence of bleeding (≥1 site or line/profuse bleeding) and/or suppuration on gentle probing around the implant
* Systemically healthy adults
* Able to provide written informed consent

Exclusion Criteria:

* Use of anticoagulants, anti-aggregants, antibiotics, or corticosteroids in the past 3 months
* Pregnant or lactating women
* Inability to perform adequate oral hygiene

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Change in plaque score at implant sites | through study completion, an average of 3 months
  Change in plaque score at implant sites, recorded at four/six sites per implant using a standardized plaque index system.
Change in bleeding score at implant sites | through study completion, an average of 3 months
  Change in bleeding score at implant sites, recorded at four/six sites per implant using a standardized plaque index system.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUS, Siena, Italy

IPD SHARING:
Plan to Share IPD: No